CLINICAL TRIAL: NCT01336933
Title: A Phase II Study of Cyclophosphamide, Etoposide, Vincristine and Prednisone (CEOP) Alternating With Pralatrexate (P) as Front Line Therapy for Patients With Stage II, III and IV Peripheral T-Cell Non-Hodgkin Lymphoma
Brief Title: Combination Chemotherapy and Pralatrexate as First-Line Therapy in Treating Patients With Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0569-10-FB; NCI-2011-00254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2011-03-23; First posted 2011-04-18 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Hepatosplenic T-cell Lymphoma; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Peripheral | interventions — Prednisone; Cyclophosphamide; Etoposide; Vincristine; 10-propargyl-10-deazaaminopterin; Comparative Genomic Hybridization; Gene Expression Profiling; Base Sequence; Immunohistochemistry; Microarray Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): "A" Treatment: Cyclophosphamide,Etoposide, Vincristine and Prednisone (CEOP) "B" Treatment: Pralatrexate (P)
  "A" cycles (CEOP) of the treatment regimen are 14 days, followed by " B" cycles (P) which are 21 days, followed by 7 days of rest for a total of 42 days per course, unless criteria are met for stopping or holding treatment or to a maximum of 6 courses.
  Patients with Complete Response (CR) or Partial Response (PR), per investigators discretion, may then undergo hematopoietic stem cell collection and administration of standard preparative regimen followed by hematopoietic stem cell transplantation.
  Interventions: Drug: prednisone; Drug: cyclophosphamide; Drug: etoposide; Drug: Vincristine; Drug: pralatrexate; Other: laboratory biomarker analysis; Genetic: comparative genomic hybridization; Genetic: gene expression analysis; Genetic: nucleic acid sequencing; Genetic: mutation analysis; Other: immunohistochemistry staining method; Genetic: microarray analysis; Genetic: RNA analysis

INTERVENTIONS:
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: etoposide — Given PO or IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: Vincristine — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: pralatrexate — Given IV
  Other Names: FOLOTYN; PDX
Other: laboratory biomarker analysis — Correlative studies
Genetic: comparative genomic hybridization — Correlative studies
  Other Names: comparative genomic analysis
Genetic: gene expression analysis — Correlative studies
Genetic: nucleic acid sequencing — Correlative studies
  Other Names: Gene Sequencing; Molecular Biology, Nucleic Acid Sequencing
Genetic: mutation analysis — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: microarray analysis — Correlative studies
  Other Names: gene expression profiling
Genetic: RNA analysis — Correlative studies

SUMMARY:
This phase II trial studies how well combination chemotherapy and pralatrexate works in treating patients with non-Hodgkin lymphoma (NHL). Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate in a Phase II study a preliminary estimate of the complete response (CR) rate of a new chemotherapy regimen involving Cyclophosphamide, Etoposide, Vincristine and Prednisone (CEOP) alternating with Pralatrexate (P) as front line therapy for patients with Stage II, III and IV Peripheral T-Cell NHL not otherwise specified (NOS), Anaplastic large cell lymphoma (ALK negative), Angioimmunoblastic T-cell lymphoma, Enteropathy associated T-cell lymphoma, Hepatosplenic gamma delta T-cell lymphoma followed by an optional stem cell transplant with high dose chemotherapy and Autologous stem cell transplant.

SECONDARY OBJECTIVES:

I. To evaluate partial response (PR). II. To evaluate overall response (CR+PR). III. To evaluate the safety and tolerability of the regimen IV. To assess the 2 year event free survival (EFS) and overall survival (OS) using this regimen.

V. To assess the percentage of patients who proceeded with transplant. VI. To evaluate the ability to collect peripheral blood stem cells after this regimen.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) and vincristine IV on day 1, etoposide IV on days 1-3 or orally (PO) once daily (QD) on days 2-3, and prednisone PO QD on days 1-5 (CEOP administration). Patients also receive pralatrexate IV over 3-5 minutes on days 15, 22, and 29 (P administration). Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients with Complete Response (CR) or Partial Response (PR), per investigators discretion, may then undergo hematopoietic stem cell collection and administration of standard preparative regimen followed by hematopoietic stem cell transplantation.

After completion of study treatment, patients are followed up for 2 years (transplant patients) or periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed new diagnosis of Stage II, III and IV peripheral T-cell NHL not otherwise specified (NOS), anaplastic large cell lymphoma (ALK negative) (ALK positive if international prognostic index [IPI] 3, 4, or 5), angioimmunoblastic T-cell lymphoma, enteropathy associated T-cell lymphoma, hepatosplenic gamma delta T-cell lymphoma
* Pathology material (hematoxylin and eosin [H&E] stain, immunohistochemistry [IHC] and pathology report from initial diagnosis, if slides are not available, then 8 unstained slides of 4 micron thickness or a representative block should be sent) will be reviewed, and the diagnosis confirmed by University Nebraska Medical Center (UNMC) pathology department (retrospective diagnostic review: treatment may commence prior to the UNMC review)
* No prior therapy with the exception of prior radiation therapy and 1 cycle of chemotherapy based on current diagnosis and clinical condition
* Age 19 years or older (the age of consent in Nebraska); age 18 years or older (applicable to states where the age of majority is 18)
* Expected survival duration of >= six months
* Karnofsky Performance Status >= 70
* Absolute neutrophil count (ANC) >= 1000 cells/mm^3, unless due to lymphoma involvement of the bone marrow
* Platelet Count >= 100 mm^3, unless due to lymphoma involvement of the bone marrow
* Total bilirubin =< 1.5 x upper normal limit (ULN), or =< 3 x ULN if documented hepatic involvement with lymphoma, or =< 5 x ULN if history of Gilbert's Disease
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (=< 5 x ULN if documented hepatic involvement with lymphoma)
* Serum potassium within normal range
* Serum creatinine < 2.0 mg/dL or calculated creatinine clearance (CrCl) > 45 mL/min
* Prothrombin time (PT) or international normalized ratio (INR), and partial thromboplastin time (PTT) =< 1.5 x ULN unless patient is receiving anticoagulants; if patient is on anticoagulation therapy, levels should be within therapeutic range
* Patients with measurable disease; patients with non-measurable but evaluable disease may be eligible after discussion with the principal investigator (PI); baseline measurements and evaluations must be obtained within 6 weeks of registration to the study; abnormal positron emission tomography (PET) scans will not constitute evaluable disease, unless verified by computed tomography (CT) scan or other appropriate imaging
* Patients with measurable disease must have at least one objective measurable disease parameter; a clearly defined, bidimensionally measurable defect or mass measuring at least 2 cm in diameter on a CT scan will constitute measurable disease; proof of lymphoma in the liver is required by a confirmation biopsy
* Women must not be pregnant or breast-feeding due to teratogenic effects of chemotherapy

  * All females of childbearing potential must have a blood test within 2 weeks prior to registration to rule out pregnancy
  * Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Male and female patients of reproductive potential must agree follow accepted birth control measures
* Patient must be able to adhere to the study visit schedule and other protocol requirements
* Patients must be willing to give written informed consent, and sign an institutionally approved consent form before performance of any study-related procedure not part of normal medical care; with the exception of 1 cycle of chemotherapy based on current diagnosis and clinical condition, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* No serious disease or condition that, in the opinion of the investigator, would compromise the patient's ability to participate in the study

Exclusion Criteria:

* Pregnant or breast feeding females
* Known positive for human immunodeficiency virus (HIV), human T-lymphotropic virus type 1 (HTLV-1), or infectious hepatitis, type A, B or C or active hepatitis
* Major surgery within 2 weeks of study drug administration
* Prior malignancies within the past 3 years with exception of adequately treated basal cell, squamous cell skin cancer, or thyroid cancer; carcinoma in situ of the cervix or breast; prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen (PSA) levels
* Patients with a diagnosis of other peripheral T-cell lymphoma (PTCL) histologies other than those specified in the inclusion criteria
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* Concomitant administration of nonsteroidal anti-inflammatory drugs (NSAIDs) and trimethoprim/sulfamethoxazole will not be allowed, since these may result in delayed clearance of pralatrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, Principal Investigator — University of Nebraska
Locations (9):
- United States (9):
  - Mayo Clinic, Arizona, Scottsdale, Arizona
  - Stanford University, Stanford, California
  - Emory University School Of Medicine, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center, Washington University, St Louis, Missouri
  - Eppley Cancer Center, University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Advani RH, Ansell SM, Lechowicz MJ, Beaven AW, Loberiza F, Carson KR, Evens AM, Foss F, Horwitz S, Pro B, Pinter-Brown LC, Smith SM, Shustov AR, Savage KJ, Vose JM. A phase II study of cyclophosphamide, etoposide, vincristine and prednisone (CEOP) Alternating with Pralatrexate (P) as front line therapy for patients with peripheral T-cell lymphoma (PTCL): final results from the T- cell consortium trial. Br J Haematol. 2016 Feb;172(4):535-44. doi: 10.1111/bjh.13855. Epub 2015 Dec 2. PMID 26627450

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy and Enzyme Inhibitor Therapy: "A" Treatment: Cyclophosphamide,Etoposide, Vincristine and Prednisone (CEOP) "B" Treatment: Pralatrexate (P)
  "A" cycles (CEOP) of the treatment regimen are 14 days, followed by " B" cycles (P) which are 21 days, followed by 7 days of rest for a total of 42 days per course, unless criteria are met for stopping or holding treatment or to a maximum of 6 courses.
  Patients with Complete Response (CR) or Partial Response (PR), per investigators discretion, may then undergo hematopoietic stem cell collection and administration of standard preparative regimen followed by hematopoietic stem cell transplantation.
Period: Overall Study
Arm/Group | Chemotherapy and Enzyme Inhibitor Therapy
Started | 34
Completed | 33
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Chemotherapy and Enzyme Inhibitor Therapy): Cyclophosphamide and vincristine sulfate by IV on day 1, etoposide IV on days 1-3 or by mouth (PO), once a day (QD) on days 2-3, and prednisone PO QD on days 1-5 (CEOP administration). Patients also receive pralatrexate IV over 3-5 minutes on days 15, 22, and 29 (P administration). Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients with CR or PR, per investigators discretion, may then undergo hematopoietic stem cell collection and administration of standard preparative regimen followed by hematopoietic stem cell transplantation.
  prednisone: Given PO
  cyclophosphamide: Given IV
  etoposide: Given PO or IV
  vincristine sulfate: Given IV
  pralatrexate: Given IV
  laboratory biomarker analysis: Correlative studies
  comparative genomic hybridization: Correlative studies
  gene expression analysis: Correlative studies
  nucleic acid sequencing: Correlative studies
  mutation analysis
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 62 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate of Cyclophosphamide, Etoposide, Vincristine and Prednisone (CEOP) and Pralatrexate (P) Treatment
Description: Complete Response Rate (CR) was reported at the end of the CEOP-P (6 courses for patients not receiving transplant and 4-6 courses for patients receiving transplant). Response assessment was performed by computerized tomography (CT) or positron emission tomography (PET)/CT based on the investigator's preference after cycles 2, 4 and 6. Response was assessed by the treating physician according to the Cheson Revised response criteria (Cheson et al,, 2007) or International Harmonization Project criteria (Cheson, 2007), based on imaging modality used.
  Complete Response Definition: Disappearance of all evidence of disease Nodal Masses: (a) [18F]fluorodeoxyglucose(FDG)-avid or PET positive prior to therapy; mass of any size permitted if PETnegative (b) Variably FDG-avid or PET negative; regression to normal size on CT Spleen, Liver: Not palpable, nodules disappeared Bone Marrow: Infiltrate cleared on repeat biopsy; if indeterminate by morphology, immunohistochemistry should be negative
Time Frame: 168 days - 252 days (4-6 courses; 42 days per course)
Measure: Number; unit: percentage of participants analyzed
Groups:
- Treatment (Chemotherapy and Enzyme Inhibitor Therapy): Patients receive cyclophosphamide IV and vincristine sulfate IV on day 1, etoposide IV on days 1-3 or PO QD on days 2-3, and prednisone PO QD on days 1-5 (CEOP administration). Patients also receive pralatrexate IV over 3-5 minutes on days 15, 22, and 29 (P administration). Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients with CR or PR, per investigators discretion, may then undergo hematopoietic stem cell collection and administration of standard preparative regimen followed by hematopoietic stem cell transplantation.
  prednisone: Given PO
  cyclophosphamide: Given IV
  etoposide: Given PO or IV
  vincristine sulfate: Given IV
  pralatrexate: Given IV
  laboratory biomarker analysis: Correlative studies
  comparative genomic hybridization: Correlative studies
  gene expression analysis: Correlative studies
  nucleic acid sequencing: Correlative studies
  mutation analysis: Correlative studies
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 33
percentage of participants analyzed | 52

2. Secondary Outcome: Overall Response Rates (ORR)= (Complete Response Rates (CR) + Partial Response Rates (PR))
Description: Every patient who fulfills all aspects of patient eligibility who receives at least 2 complete courses of chemotherapy will be evaluable for the response endpoint. Response rates will be descriptively summarized using percentages and 95% confidence intervals.
  Complete Response Definition: Defined in Primary Objective Partial Response Definition: Regression of measurable disease and no new sites, Nodal Masses: > 50% decrease in sum of the product of the diameters (SPD) of up to 6 largest dominant masses; no increase in size of other nodes
  1. FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site
  2. Variably FDG-avid or PET negative; regression on CT Spleen, Liver:> 50% decrease in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen Bone Marrow: Irrelevant if positive prior to therapy; cell type should be specified
Time Frame: 2 years
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 33
percentage of participants analyzed | 70

3. Secondary Outcome: Event Free Survival (EFS)
Description: Estimated 2-year Event Free Survival (EFS), as well as plots of EFS, will be produced using the method of Kaplan-Meier, along with 95% confidence intervals for EFS. Event-free survival is defined as time from therapy until relapse, progression, or death from any cause.
Time Frame: 2 years
Population: All evaluable patients irrespective of the total number of cycles of therapy received were included in the EFS and OS analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants analyzed
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 33
percentage of participants analyzed | 39 [21 to 57]

4. Secondary Outcome: Overall Survival (OS)
Description: Estimated 2-year Overall Survival (OS), as well as plots of OS, will be produced using the method of Kaplan-Meier, along with 95% confidence intervals for OS. Overall survival is defined as time from the first chemotherapy administered on trial until death from any cause.
Time Frame: 2 years
Population: All evaluable patients irrespective of the total number of cycles of therapy received were included in EFS and OS analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants analyzed
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 33
percentage of participants analyzed | 60 [39 to 76]

5. Secondary Outcome: To Evaluate the Safety and Tolerability of the Regimen by the Percent of Participants With Indicated Adverse Events
Description: Adverse events will be summarized using patient level incidence rates so that a patient contributes once to any adverse event. The number and percentage of patients with any adverse event will be summarized for each course. Serious adverse events will be analyzed similarly.
Time Frame: 22 months
Population: All eligible patients who received at least one cycle of chemotherapy were evaluable for toxicity.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 33
percentage of participants
  Grade 3-4 anaemia | 27
  Grade 3-4 thrombocoytopenia | 12
  Grade 3-4 febrile neutropenia | 18
  Grade 3-4 mucositis | 18
  Grade 3-4 sepsis | 15
  Grade 3-4 increased creatinine | 12
  Grade 3-4 liver transaminases | 12

6. Secondary Outcome: Percent of Patients Who Proceeded With Transplant
Description: Percentage of patients who received consolidation with high dose therapy and autologous stem cell rescue (HDT/SCR).
Time Frame: 168-252 days (4 courses up to 6 courses of treatment)
Population: Thirty-three patients were analyzed. One patient withdrew consent before starting therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 33
Participants | 15

ADVERSE EVENTS:
Time Frame: 20 months
Description: Adverse Event Reporting: Grade 3 and greater using the CTCAE coding (4.0)
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor Therapy)
All-Cause Mortality (participants affected / at risk) | 12/33
Serious Adverse Events (participants affected / at risk) | 13/33
Other Adverse Events (participants affected / at risk) | 19/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Enzyme Inhibitor Therapy) (N=33)
Fever (General disorders) | 4 (6)
Lung Infection (Infections and infestations) | 3 (4)
Headache (Nervous system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Sepsis (Infections and infestations) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — cellulitis
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Acute respiratory distress syndrome (ARDS)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Kidney anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Hypoxia (Reproductive system and breast disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Cardiac disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Creatinine increased
Agitation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Enzyme Inhibitor Therapy) (N=33)
Neutrophil count decreased (Investigations) | 7 (9)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (5) — decreased leukocytes
Anemia (Blood and lymphatic system disorders) | 7 (14)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Creatinine increased (Investigations) | 3 (4)
Fever (General disorders) | 3 (3)
hypocalcemia (Metabolism and nutrition disorders) | 3 (7)
White blood cell decreased (Investigations) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No